CLINICAL TRIAL: NCT03084601
Title: Evaluation of Postoperative Pain After Using 3MIX-TATIN Versus Calcium Hydroxide Iodoform Paste In Necrotic Primary Molars Treated by Lesion Sterilization and Tissue Repair Therapy: A Randomized Controlled Trial
Brief Title: Evaluation of Postoperative Pain After Using 3MIX-TATIN Versus Calcium Hydroxide Iodoform Paste In Necrotic Primary Molars Treated by Lesion Sterilization and Tissue Repair Therapy
Acronym: 3-mixtatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahmoud M Saadoon (Other)
Responsible Party: Sponsor-Investigator, Mahmoud M Saadoon, resident dr, department of pedodontics, cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mahmoud 3-mixtatin
Record Dates: First submitted 2017-02-13; First posted 2017-03-21 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Necrotic Pulp; Postoperative Pain
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative | interventions — Calcium Hydroxide; iodoform; Ointments; Metapex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium hydroxide iodoform paste (Active Comparator): intervention administered to control group is a combination of drugs as follow: ciprofloxacin 500mg, cefixime 500 mg, metronidazole 500 mg, simvastain 40mg. all are mixed, placed in pulp chamber only one time and tooth is restored
  Interventions: Drug: 3-mixtatin
- 3-mixtatin (Experimental): intervention administered to experimental group is a ready made mixture of calcium hydroxide and iodoform, placed in pulp chamber only one time and tooth is restored
  Interventions: Drug: Calcium Hydroxide, Iodoform, paste

INTERVENTIONS:
Drug: Calcium Hydroxide, Iodoform, paste — mixture of calcium hydroxide and iodoform
  Other Names: metapex
  Arms: 3-mixtatin
Drug: 3-mixtatin — 3-mixtatin mixture of ciprofloxacin, metronidazole, cefixime, and simvastatin
  Other Names: 3mixtatin
  Arms: calcium hydroxide iodoform paste

SUMMARY:
The aim of the current study is to compare a newly introduced material which is a combination of triple mix antibiotics paste and anti-hyperlipidemia drug simvastatin, the new material is named 3MIX-TATIN & will be compared to triple antibiotic paste for management of necrotic primary molars by using lesion sterilization and tissue repair LSTR technique.

DETAILED DESCRIPTION:
3Mix-tatin will prepared by mixing three commercially available antibiotics with simvastatin. After removing the coating materials, 3 types of antibiotics are pulverized by porcelain mortars and pestles to achieve fine powders. A total of 100 mg ciprofloxacin, 100 mg metronidazole, and 100 mg cefixime will be mixed in a ratio of 1: 1: 1. Two milligrams of simvastatin will be added to the drugs blend to form 3-Mix-tatin. Preparation of 3Mixtatin will be trained and supervised by an expert pharmacist. 3Mixtatin will be stored in a tightly capped porcelain container, adding a small amount of silica gel in a bag inside the container to maintain low humidity. This powder will be mixed with normal saline to form a creamy paste of 3Mixtatin at the time of application.

Local anesthesia using mepivicaine hydrochloride 3% (septodont, saint-maurdesFosses, France) will be administered.

Rubber dam isolation.

Access cavity will be prepared with a fissure bur in a high-speed handpiece, necrotic pulp tissue will be removed using a sterile sharp spoon excavator.

The canal orifices will be enlarged with a round bur (one mm diameter and two mm depth) to create medication receptacles.

Cotton pellet moistened with 2.5% sodium hypochlorite (NaOCl) will be placed in the pulp chamber for 1 minute.

Bleeding, if present, will be controlled by applying sterile cotton pellet moistened with 10% sodium hypochlorite against the pulp stumps and will be maintained for 1 min.

The 3-Mix-Tatin will be mixed with saline to obtain a creamy mix and placed over the canal orifices and the pulpal floor.

The access opening will be sealed with a glass ionomer cement , and the tooth will be restored with a stainless steel crown.

ELIGIBILITY:
Inclusion Criteria:

* Children age range from 5-8 years.
* Children free from any systemic diseases or medical problems.
* Primary molar with necrotic pulp, with pain, gingival abscess, fistula openings, or clinical mobility not exceeding grade two.
* Radiographic evidence of non-perforating internal resorption, external resorption not exceeding 1\3 of the root, furcation or periapical radiolucency.

Exclusion criteria:

* Non-restorable molars or beyond repair, for example: decay reaches to bifurcation, a hard gingival margin cannot be established or infection cannot be eradicated by other mean (Balaji, 2007).
* Patient with known allergy to any type of antibiotics or anti-hyperlipidemia drugs.
* Patient with facial cellulitis or lymphadenopathy
* Lack of patient/parent compliance and cooperation.
* Refusal of participation or failure to obtain an informed consent.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
pain | at 3rd months
  measurment of post-operative pain by a questionnaire either present or absent

SECONDARY OUTCOMES:
swelling | at 3rd month
  visual inspection either present or absent
swelling | at 6th month
  visual inspection either present or absent
swelling | at 9th month
  visual inspection either present or absent
mobility | at 3rd month
  visual inspection either present or absent
mobility | at 6th month
  visual inspection either present or absent
mobility | at 9th month
  visual inspection either present or absent

CONTACTS AND LOCATIONS:
Locations (1):
- Pedodontic Department Cairo University, Cairo Governorate, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No